CLINICAL TRIAL: NCT01177709
Title: Evaluation of the Efficacy of Metformin for Weight Loss and Metabolic Effects In Overweight Psychiatric Patients Treated With Antipsychotic Medication
Brief Title: Metformin for Weight Loss in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moved to different institution. Decided to concentrate on different studies.
Sponsor: Nathan Kline Institute for Psychiatric Research (Other)
Responsible Party: Principal Investigator, Robert C. Smith MD PhD, Research Psychiatrist-Principal investigator, Nathan Kline Institute for Psychiatric Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 091/C22
Record Dates: First submitted 2010-04-23; First posted 2010-08-09 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Schizophrenia; Obesity
Keywords: schizophrenia; antipsychotics; obesity; diabetes
MeSH Terms: conditions — Schizophrenia; Obesity; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — metformin 500- 2500 mg/day. Patient received variable doses of metformin starting at 500 mg/day and increasing up to maximum of 2500 mg/day over 3-4 weeks. Dose was titrated on tolerability and side effects, especially development of hypoglycemia. This explains why different patients received different maximum doses.

SUMMARY:
Study hypothesis is that patients on antipsychotics medication treated with metformin will show loss in weight and improved measures of glucose metabolism.

DETAILED DESCRIPTION:
Patients who had gained more than 10 lbs of weight in the last 3 months or had BMI of 35 or greater were treated with metformin up to 2500 mg/day in an open label study of up to 3 months time. Changes in weight and glucose measures were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be 18-70 years of age;
* Currently hospitalized or an outpatient at MPC;
* BMI ≥ 35 or excessive recent weight gain ( > than 10 lb weight gain in the past 3 months);
* Patients will have a diagnosis of schizophrenia or schizoaffective disorder or bipolar disorder.

Exclusion Criteria:

* Age below 18 or over 70;
* Patient is currently already treated with metformin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Smith, MD PHD, Principal Investigator — Nathan Kline Institute for Psychiatric Research
Locations (1):
- Manhatan Psychiatric Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin: Metformin: metformin 500- 2500 mg/day.
Period: Overall Study
Arm/Group | Metformin
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Weight (wt) in Pounds (Lbs)..
Description: Patients weight in pounds
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Mean (Standard Error); unit: weight(wt) in pounds(lbs)
Arm/Group | Metformin
Number analyzed (Participants) | 12
weight(wt) in pounds(lbs)
  baseline wt lbs | 250.97 (11.52)
  4 week wt lbs | 244.73 (10.84)
  8 week wt lbs | 244.15 (10.06)
  12 week wt lbs | 240.44 (9.22)

2. Secondary Outcome: Glucose Levels
Description: Fasting glucose
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Metformin
Number analyzed (Participants) | 12
mg/dL
  basline glucose | 111.05 (12.83)
  week 4 glucose | 87.00 (2.95)
  week 8 glucose | 89.17 (2.17)
  week 12 gluocse | 94.25 (3.85)

3. Secondary Outcome: Insulin Level
Description: fasting serum insulin uIU/ml.
Time Frame: baseline, 4 weks, 8 weeks, 12 weeks
Measure: Mean (Standard Error); unit: uIU/ml
Arm/Group | Metformin
Number analyzed (Participants) | 12
uIU/ml
  baseline insulin | 11.18 (1.32)
  week 4 insulin | 11.53 (21.71)
  week 8 insulin | 8.85 (1.41)
  week 12 insulin | 11.29 (2.39)

ADVERSE EVENTS:
Arm/Group | Metformin
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=12)
low serum sodium, (Renal and urinary disorders) | 1 (1) — patient developed low serum sodium while on additional medication chlorothiazide for kidney problems
penumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — patient developed pneumonia after the study was completed; not related to study drug.

LIMITATIONS AND CAVEATS:
This is an open non-blinded study in a small number of subjects. However, it is unlikely that outcomes measures of weight, glucose, and insulin, would have been likely to be affected by non-blinding of subjects and investigators. .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No